CLINICAL TRIAL: NCT05483361
Title: Effect Of Smart Phone Addiction On Pulmonary Function, And Functional Capacity In Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Mohamed Abd Elrazek Eletreby, assistant lecturer, Cairo University
Other Study IDs: P.T.REC/012/003600
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Smartphone Addiction; Pulmonary Function; Functional Capacity; School Age Children
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smart phone addiction group: Smart phone addiction will be assessed using the Smart Phone Addiction Scale short version (SAS-SV) evaluation of pulmonary functions and functional capacity evaluation craniovertebral angle

SUMMARY:
Statement of the problem:

Are there relations between smartphone addiction, neck posture, pulmonary functions and functional capacity in children? Null hypothesis

It will be assumed that:

* There will be no effect of smart phone addiction on head posture, pulmonary function and functional capacity in children.
* There will be no relation between smartphone addiction, head posture, pulmonary function and functional capacity in children.

DETAILED DESCRIPTION:
Subjects:

Sample size estimation will be carried out to determine the recruited number of children selected randomly from both governmental and private primary and preparatory schools at El Mansoura educational administration, Dakahlia Governorate and Damietta governorate to participate in this study. The survey targets the normal students from both sexes.

They will be selected based on the following:

Inclusion criteria:

* All children will be age ranges from 10 to 12 years
* The BMI <95th percentile (WHO, 2007)
* Smartphone addiction scale short version will be used to categorize the children to addicted group (score > 32) (Kwon et al., 2013) .
* They will be cooperative and followed the instructions.

Exclusive criteria:

Children will be excluded from the study if they have:

* Neurological diseases.
* Respiratory disorders.
* Congenital deformities.
* Vision disorders not corrected by glasses.
* Children who participate in competitive sports.
* Obesity.

ELIGIBILITY:
Inclusion Criteria:

* All children will be age ranges from 10 to 12 years
* The BMI <95th percentile (WHO, 2007)
* Smartphone addiction scale short version will be used to categorize the children to addicted group (score > 32) (Kwon et al., 2013) .
* They will be cooperative and followed the instructions.

Exclusion Criteria:

* • Neurological diseases.

  * Respiratory disorders.
  * Congenital deformities.
  * Vision disorders not corrected by glasses.
  * Children who participate in competitive sports.
  * Obesity.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of pulmonary functions | baseline only
  Computerized spirometer is the most frequently used measure of lung function and is a measure of volume against time. It is a simple and quick procedure to perform

SECONDARY OUTCOMES:
evaluation of functional capacity | baseline only
  By 3 minutes step test It is based on the principles that your heart rate will return to normal quickly the fitter you are the value of post- exercise heart is considered to be an indicator to cardiovascular fitness

OTHER OUTCOMES:
evaluation craniovertebral angle | baseline only
  By Kinovea computer program A free 2D motion analysis software

CONTACTS AND LOCATIONS:
Overall Officials: yasmine eletreby, Principal Investigator — Cairo University
Locations (1):
- Governmental and Private Primary and Preparatory Schools, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided